CLINICAL TRIAL: NCT05013866
Title: Repair of Proximal Restoration With Resin Composite Bulk-Fill. Double Blind Randomized Clinical Trial
Brief Title: Repair of Proximal Restoration Resin Bulk Fill. Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Patricio Vildosola Grez, Clinical Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIFO 2017/001
Record Dates: First submitted 2021-08-04; First posted 2021-08-19 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Dental Diseases
Keywords: Composite Dental Resin
MeSH Terms: conditions — Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repair of resin Z350 (Active Comparator): Repair with Z350 on resin composite proximal
  Interventions: Procedure: Repair resin composite proximal
- Repair of Tetric Evo Ceram Bulkfill (Experimental): Repair with Tetric Evo Ceram on resin composite proximal
  Interventions: Procedure: Repair resin composite proximal

INTERVENTIONS:
Procedure: Repair resin composite proximal — Repair proximal composite resin restoration, removing the defective material and then restoring it with another composite resin

SUMMARY:
Bulk Fill" (RBF) composite resins (RC) has been on the market, with the main advantage of being applied in a single layer, faster and easier than a conventional RC. Repair of RC restorations is a validated treatment option in dentistry, which has been shown to increase the longevity of restorations by minimizing tooth damage such as complete replacement. Currently there are no clinical studies that support the actual performance of RBF repair

DETAILED DESCRIPTION:
Main objective: Compare the clinical performance with FDI of repairs proximal RC restorations between a conventional resin and a RBF in a period of 24 months. Hypothesis: There is not different clinical performance of proximal RC repairs done with RBF when compared to conventional RC repairs. Material and method: 80 volunteer patients will be randomly recruited to attend the clinic of the Faculty of Dentistry of the University of Chile who have two proximal RC restorations with indication of repair according to the FDI system (n per group = 80). Each patient must accept and sign an informed consent. The repairs will be randomly divided into two groups on the same patient. Control Group: Conventional RC repair (Z350 XT). Experimental Group: RBF (Tetric Evoceram Bulk Fill) Repair. For the restorative technique, a three-step adhesive with acid-etched enamel-dentin will be used. It will be evaluated at 2 weeks (Baseline), at 6, 12, 18, 24 months by two blind and calibrated evaluators (Cohen Kappa> 0.8). The data will be analyzed with the SSPS 21.0 software and the Friedman, Wilcoxon and Mann Whitney tests will be applied with a significance level of 95%.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years,
* healthy
* high cariogenic risk,
* Vital molars and premolars,
* Natural antagonist and proximal
* Indication of repair in the proximal with depth> 2mm.

Exclusion Criteria:

* Patients has xerostomia either by taking medications known to produce xerostomia or those with radiation induced or Sjogren's syndrome patients -inability to perform hygiene
* pregnant women
* severe bruxism
* Prosthesis
* Not absolute isolation
* Tooth fracture and / or restoration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical Performance | Baseline
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI System, Unit is Ranking system has 5 scores for each different property. Either restoration is clinically excellent (1), or good (2), or sufficient(3), or unsatisfactory(4), or clinically poor(5).
Clinical Performance | 12 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI System, Unit is Ranking system has 5 scores for each different property. Either restoration is clinically excellent (1), or good (2), or sufficient(3), or unsatisfactory(4), or clinically poor(5).
Clinical Performance | 18 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI System, Unit is Ranking system has 5 scores for each different property. Either restoration is clinically excellent (1), or good (2), or sufficient(3), or unsatisfactory(4), or clinically poor(5).
Clinical Performance | 24 months
  Outcome measure is Clinical performance of composite resin restoration, Device for measurement is FDI System, Unit is Ranking system has 5 scores for each different property. Either restoration is clinically excellent (1), or good (2), or sufficient(3), or unsatisfactory(4), or clinically poor(5).

CONTACTS AND LOCATIONS:
Overall Officials: Patricio Vildosola, Principal Investigator — University of Chile
Locations (1):
- Patricio Vildosola Grez, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No